CLINICAL TRIAL: NCT00769483
Title: A Phase I/ Randomized Phase II Study of Gemcitabine Plus Erlotinib Plus MK-0646; Gemcitabine Plus MK-0646 and Gemcitabine Plus Erlotinib for Patients With Advanced Pancreatic Cancer (IISP#33337)
Brief Title: MK-0646 and Gemcitabine +/- Erlotinib for Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0910; NCI-2010-01049 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Results first posted 2019-03-20 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Pancreatic Cancer; Pancreatic Adenocarcinoma
Keywords: Pancreas; Pancreatic Cancer; Advanced cancer of the pancreas; Pancreatic Adenocarcinoma; MK-0646; Gemcitabine; Gemzar; Erlotinib hydrochloride; Erlotinib; OSI-774; Tarceva
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — dalotuzumab; Gemcitabine; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Phase I, Arm A (Experimental): MK-0646 + Gemcitabine
  Interventions: Drug: MK-0646; Drug: Gemcitabine
- Phase I, Arm B (Experimental): MK-0646 + Gemcitabine + Erlotinib
  Interventions: Drug: MK-0646; Drug: Gemcitabine; Drug: Erlotinib
- Phase II, Arm A (Experimental): Gemcitabine + Erlotinib
  Interventions: Drug: MK-0646; Drug: Gemcitabine
- Phase II, Arm B (Experimental): MK-0646 + Gemcitabine + Erlotinib
  Interventions: Drug: MK-0646; Drug: Gemcitabine; Drug: Erlotinib
- Phase II, Arm C (Experimental): Gemcitabine + Erlotinib
  Interventions: Drug: Gemcitabine; Drug: Erlotinib

INTERVENTIONS:
Drug: MK-0646 — Starting Dose Level: 5 mg/kg given intravenously over 60 minutes Days 1, 8, 15, 22 of 28 Day Cycle.
  Arms: Phase I, Arm A; Phase I, Arm B; Phase II, Arm A; Phase II, Arm B
Drug: Gemcitabine — 1000 mg/m^2 given intravenously over 1-1/2 hours Days 1, 8, and 15 of each 28 Day Cycle.
  Other Names: Gemzar; Gemcitabine Hydrochloride
Drug: Erlotinib — 100 mg by mouth daily.
  Other Names: OSI-774; Tarceva; Erlotinib Hydrochloride
  Arms: Phase I, Arm B; Phase II, Arm B; Phase II, Arm C

SUMMARY:
Objectives:

Primary Objectives:

* Phase I: Determine the maximal tolerated dose (MTD) of MK-0646 in combination with gemcitabine or gemcitabine plus erlotinib and recommended phase II dose.
* Phase II:

  * Assess progression-free survival (PFS) with a) gemcitabine plus MK-0646 b) gemcitabine plus erlotinib plus MK-0646 and c) gemcitabine plus erlotinib.
  * Explore IGF1 tissue level as a predictive biomarker for MK-0646 therapy in phase II expansion cohort.

Secondary Objectives:

* Assess overall response rate (ORR), treatment toxicity, and overall survival (OS) with the addition of MK-0646 to gemcitabine or gemcitabine plus erlotinib.
* Correlate PFS and OS with IGF-1, IGFBP-3 levels and the expression of p-IRS, IGF-1R, EMT biomarkers, Akt, Erk, mTOR, and PI13k in tumor cells.
* To assess the incidence of single nucleotide polymorphisms of the IgF1R pathway related genes (IGF1, IGF1R, IRS1 and IRS2). These genotypes will be correlated with the clinical endpoints of this study, including OS, ORR and PFS.

DETAILED DESCRIPTION:
Phase I

The Study Drugs:

MK-0646 is designed to block proteins that are thought to cause cancer cells to grow and spread. This drug may help slow the growth of tumors.

Gemcitabine is designed to disrupt the growth of cancer cells, which may cause cancer cells to die.

Erlotinib hydrochloride is designed to block the activity of a protein found on the surface of many tumor cells that may control the growth and survival of cancer cells. This may stop cancer cells from growing.

Study Drug Dose Level and Groups:

If you are found to be eligible to take part in this study, you will be assigned to a group (Arm A or Arm B) based on when you joined the study, how many participants have been enrolled before you, and on the safety data that is available at that time.

* If you are in Arm A, you will receive MK-0646 and gemcitabine.
* If you are in Arm B, you will receive MK-0646, gemcitabine, and erlotinib hydrochloride.

There are 2 dose levels of MK-0646 in each arm. There will be 3-6 participants enrolled in each dose level in each arm. Enrollment will begin in Arm A. Arm B will use the same 2 dose levels as Arm A. If the first dose level of Arm A is found to be tolerable, at least 3 patients will be enrolled in Arm B, Level 1, and then at least 3 patients will be enrolled in Arm A, Level 2. If Arm B, Level 1 and Arm A, Level 2 can be safely given, the last group of 3-6 patients will be enrolled in Arm B, Level 2. The first group of participants in each arm will receive the lower dose level. The next group in each arm will receive a higher dose than the first group, if no intolerable side effects were seen.

The dose of gemcitabine and/or erlotinib hydrochloride will be the same for every group.

Study Drug Administration:

If you are in Arm A, on Days 1, 8, and 15 of each 28-day study cycle, you will receive gemcitabine through a needle into your vein over about 1 1/2 hours. On Days 1, 8, 15, and 22 of each cycle, you will receive MK-0646 by vein over 1 hour.

If you are in Arm B, you will take erlotinib hydrochloride by mouth once a day (in the morning) every day. You should take it with about 1 cup (8 oz.) of water 1 hour before or 2 hours after eating. On Days 1, 8, and 15 of each cycle, you will receive gemcitabine by vein over about 1 1/2 hours. On Days 1, 8, 15, and 22 of each cycle, you will receive MK-0646 by vein over 1 hour.

Depending upon how well you tolerate gemcitabine, your doctor may decide that you should receive gemcitabine on Days 1 and 15 instead of Days 1, 8, and 15.

Study Visits:

On Day 1 of Cycle 1, the following tests and procedures will be performed:

* Your medical history will be recorded.
* You will have a performance status evaluation.
* You will be asked to list any drugs you may be taking and if you have experienced any side effects.
* You will have a physical exam, including measurement of your vital signs and weight.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* Blood (about 1 teaspoon) will be drawn to make sure your body has not created cells to fight against MK-0646. These cells are called human anti-human antibodies (also known as HAHA).

On Day 8 of Cycle 1, the following tests and procedures will be performed:

* Your vital signs and weight will be measured.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will be asked if you have experienced any side effects.

On Day 15 of Cycle 1, the following tests and procedures will be performed:

* You will have a performance status evaluation.
* You will be asked to list any drugs you may be taking and if you have experienced any side effects.
* You will have a physical exam, including measurement of your vital signs and weight.
* Blood (about 2 teaspoons) will be drawn for routine tests.

On Day 22 of Cycle 1, the following tests and procedures will be performed:

* Your vital signs and weight will be measured.
* Blood (about 1 teaspoon) will be drawn to test for HAHA.
* You will be asked if you have experienced any side effects.
* Blood (about 2 teaspoons) will be drawn for routine tests.

On Day 1 of Cycles 2 and beyond, the following tests and procedures will be performed:

* You will have a performance status evaluation.
* You will be asked to list any drugs you may be taking and if you have experienced any side effects.
* You will have a physical exam, including measurement of your vital signs and weight
* Blood (about 2 teaspoons) will be drawn for routine tests.
* Blood (about 1 teaspoon) will be drawn for testing of CA 19-9.

On Days 8 and 15 of Cycles 2 and beyond, the following tests and procedures will be performed:

* Your vital signs and weight will be measured.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will be asked if you have experienced any side effects.

On Day 22 of Cycles 2 and beyond, your vital signs and weight will be measured and you will be asked if you have experienced any side effects.

On Day 22 of Cycle 2 and every even cycle (Cycles 4, 6, 8, and so on), you will have a CT scan or MRI scan to check the status of the disease. Blood (about 1 teaspoon) will also be drawn to test HAHA.

Length of Study:

You may remain on study for as long as you are benefiting. You will be taken off study if the disease gets worse or you experience intolerable side effects.

End-of-Study Visit:

After you go off study, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will have a performance status evaluation.
* You will be asked to list any drugs you may be taking and if you have experienced any side effects.
* You will have a physical exam, including measurement of your vital signs and weight.
* You will have a CT scan or MRI scan to check the status of the disease.
* Blood (about 2 teaspoons) will be collected for routine tests.
* Blood (about 1 teaspoon) will be drawn to test HAHA.
* Blood (about 1 teaspoon) will be drawn to test CA 19-9.

At Weeks 4, 8, and 12 after the end of study visit, blood (about 1 teaspoon) will be drawn to test HAHA.

Long-Term Follow Up:

Once you are off study, every 3 months from then on, the study staff will ask you how you are doing, either in the clinic or by telephone. If you are called, the phone call will take about 10-15 minutes.

This is an investigational study. MK-0646 is not FDA approved or commercially available. At this time, MK-0646 is only being used in research. Gemcitabine is FDA approved and commercially available for the treatment of pancreatic cancer. Erlotinib hydrochloride is FDA approved and commercially available for the treatment of pancreatic cancer in combination with gemcitabine.

Up to 100 patients will take part in this study. All will be enrolled at MD Anderson.

Phase II:

The Study Drugs:

MK-0646 is designed to block proteins that are thought to cause cancer cells to grow and spread. This drug may help slow the growth of tumors.

Gemcitabine is designed to disrupt the growth of cancer cells, which may cause cancer cells to die.

Erlotinib hydrochloride is designed to block the activity of a protein found on the surface of many tumor cells that may control the growth and survival of cancer cells. This may stop cancer cells from growing.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the roll of the dice) into 1 of 3 groups.

* If you are in Arm A, you will receive gemcitabine and MK-0646.
* If you are in Arm B, you will receive erlotinib hydrochloride, gemcitabine, and MK-0646.
* If you are in Arm C, you will receive erlotinib hydrochloride and gemcitabine.

Study Drug Administration:

If you are in Arm A, on Days 1, 8, and 15 of each 28-day study cycle, you will receive gemcitabine through a needle into your vein over about 1 1/2 hours as an infusion once a week for 3 weeks. On Days 1, 8, 15, and 22 of each cycle, you will receive MK-0646 by vein over 1 hour.

If you are in Arm B, you will take erlotinib hydrochloride by mouth once (in the morning) every day. On Days 1, 8, and 15 of each cycle, you will receive gemcitabine by vein over about 1 1/2 hours. On Days 1, 8, 15, and 22 of each cycle, you will receive MK-0646 by vein over 1 hour.

If you are in Arm C, you will take erlotinib hydrochloride by mouth once (in the morning) every day. On Days 1, 8, and 15 of each cycle, you will receive gemcitabine by vein over about 1 1/2 hours.

If you are taking erlotinib hydrochloride, you should take it with about 1 cup (8 oz.) of water 1 hour before or 2 hours after eating.

Depending upon how well you tolerate gemcitabine, your doctor may decide that you should receive gemcitabine on Days 1 and 15 instead of Days 1, 8, and 15.

Study Visits:

On Day 1 of Cycle 1, the following tests and procedures will be performed:

* Your medical history will be recorded.
* You will have a performance status evaluation.
* You will be asked to list any drugs you may be taking and if you have experienced any side effects.
* You will have a physical exam, including measurement of your vital signs and weight.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* If you are assigned to receive MK-0646, blood (about 1 teaspoon) will be drawn to make sure your body has not created cells to fight against MK-0646. These cells are called human anti-human antibodies (also known as HAHA).

On Day 8 of Cycle 1, the following tests and procedures will be performed:

* Your vital signs and weight will be measured.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will be asked if you have experienced any side effects.

On Day 15 of Cycle 1, the following tests and procedures will be performed:

* You will have a performance status evaluation.
* You will be asked to list any drugs you may be taking and if you have experienced any side effects.
* You will have a physical exam, including measurement of your vital signs and weight.
* Blood (about 2 teaspoons) will be drawn for routine tests.

On Day 22 of Cycle 1, the following tests and procedures will be performed if you are receiving MK-0646:

* Your vital signs and weight will be measured
* Blood (about 1 teaspoon) will be drawn to test for HAHA.
* You will be asked if you have experienced any side effects.

On Day 1 of Cycles 2 and beyond, the following tests and procedures will be performed:

* You will have a performance status evaluation.
* You will be asked about any other drugs you may be taking and if you have experienced any side effects.
* You will have a physical exam, including measurement of your vital signs and weight
* Blood (about 2 teaspoons) will be drawn for routine tests.
* Blood (about 1 teaspoon) will be drawn for testing of CA 19-9.

On Days 8 and 15 of Cycles 2 and beyond, the following tests and procedures will be performed:

* Your vital signs and weight will be measured.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will be asked if you have experienced any side effects.

On Day 22 of Cycles 2 and beyond, your vital signs and weight will be measured, (if you are receiving MK-0646). and you will be asked if you have experienced any side effects.

On Day 22 of Cycle 2 and every even cycle (Cycles 4, 6, 8, and so on), you will have a CT scan or MRI scan to check the status of the disease. Blood (about 1 teaspoon) will be also be drawn to test HAHA if you are receiving MK-0646.

Length of Study:

You may remain on study for as long as you are benefiting. You will be taken off study if the disease gets worse or you experience intolerable side effects.

If you are in Arm C (erlotinib and gemcitabine) and the disease gets worse, you may be allowed to join Arm B (gemcitabine, erlotinib, and MK-0646).

End-of-Study Visit:

After you go off study, you will have an end-of-study visit. At this visit the following tests and procedures will be performed:

* You will have a performance status evaluation.
* You will be asked to list any drugs you may be taking and if you have experienced any side effects.
* You will have a physical exam, including measurement of your vital signs and weight.
* You will have a CT scan or MRI scan to check the status of the disease.
* Blood (about 2 teaspoons) will be collected for routine tests.
* Blood (about 1 teaspoon) will be drawn for testing of CA 19-9.
* Blood (about 1 teaspoon) will be drawn for testing to test HAHA if you are receiving MK-0646.

At Weeks 4, 8, and 12 after the end of study visit, blood (about 1 teaspoon) will be drawn to test HAHA if you were receiving MK-0646.

Long-Term Follow Up:

Once you are off study, every 3 months from then on, the study staff will ask you how you are doing, either in the clinic or by telephone. If you are called, this phone call will take about 10-15 minutes.

This is an investigational study. MK-0646 is not FDA approved or commercially available. At this time, MK-0646 is only being used in research. Gemcitabine is FDA approved and commercially available for the treatment of pancreatic cancer. Erlotinib hydrochloride is FDA approved and commercially available for the treatment of pancreatic cancer in combination with gemcitabine.

Up to 100 patients will take part in this study. All will be enrolled at MD Anderson.

Phase II Expansion Cohort:

The Study Drugs:

MK-0646 is designed to block proteins that are thought to cause cancer cells to grow and spread. This drug may help slow the growth of tumors.

Gemcitabine is designed to disrupt the growth of cancer cells, which may cause cancer cells to die.

Study Treatments:

If you are found to be eligible to take part in this study, you will receive gemcitabine and MK-0646.

Study Drug Administration:

On Days 1, 8, and 15 of each 28-day study cycle, you will receive gemcitabine through a needle into your vein over about 1 1/2 hours as an infusion once a week for 3 weeks. On Days 1, 8, 15, and 22 of each cycle, you will receive MK-0646 by vein over 1 hour.

Depending upon how well you tolerate gemcitabine, your doctor may decide that you should receive gemcitabine on Days 1 and 15 instead of Days 1, 8, and 15.

Study Visits:

On Day 1 of Cycle 1, the following tests and procedures will be performed:

* Your medical history will be recorded.
* You will have a performance status evaluation.
* You will be asked to list any drugs you may be taking and if you have experienced any side effects.
* You will have a physical exam, including measurement of your vital signs and weight.
* Blood (about 2 teaspoons) will be drawn for routine tests.

On Day 8 of Cycle 1, the following tests and procedures will be performed:

* Your vital signs and weight will be measured.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will be asked if you have experienced any side effects.

On Day 15 of Cycle 1, the following tests and procedures will be performed:

* You will have a performance status evaluation.
* You will be asked to list any drugs you may be taking and if you have experienced any side effects.
* You will have a physical exam, including measurement of your vital signs and weight.
* Blood (about 2 teaspoons) will be drawn for routine tests.

On Day 22 of Cycle 1, the following tests and procedures will be performed if you are receiving MK-0646:

* Your vital signs and weight will be measured
* You will be asked if you have experienced any side effects
* Blood (about 1 tablespoon) will be drawn for biomarker testing.

On Day 1 of Cycles 2 and beyond, the following tests and procedures will be performed:

* You will have a performance status evaluation.
* You will be asked about any other drugs you may be taking and if you have experienced any side effects.
* You will have a physical exam, including measurement of your vital signs and weight
* Blood (about 2 teaspoons) will be drawn for routine tests.
* Blood (about 1 teaspoon) will be drawn for testing of CA 19-9.

On Days 8 and 15 of Cycles 2 and beyond, the following tests and procedures will be performed:

* Your vital signs and weight will be measured.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will be asked if you have experienced any side effects.

On Day 22 of Cycles 2 and beyond, your vital signs and weight will be measured and you will be asked if you have experienced any side effects.

On Day 22 of Cycle 2 and every even cycle (Cycles 4, 6, 8, and so on), you will have a CT scan or MRI scan to check the status of the disease.

Length of Study:

You may remain on study for as long as you are benefiting. You will be taken off study if the disease gets worse or you experience intolerable side effects.

End-of-Study Visit:

After you go off study, you will have an end-of-study visit. At this visit the following tests and procedures will be performed:

* You will have a performance status evaluation.
* You will be asked to list any drugs you may be taking and if you have experienced any side effects.
* You will have a physical exam, including measurement of your vital signs and weight.
* You will have a CT scan or MRI scan to check the status of the disease.
* Blood (about 2 teaspoons) will be collected for routine tests.
* Blood (about 1 teaspoon) will be drawn for testing of CA 19-9.

Long-Term Follow Up:

Once you are off study, every 3 months from then on, the study staff will ask you how you are doing, either in the clinic or by telephone. If you are called, this phone call will take about 10-15 minutes.

This is an investigational study. MK-0646 is not FDA approved or commercially available. At this time, MK-0646 is only being used in research. Gemcitabine is FDA approved and commercially available for the treatment of pancreatic cancer.

Up to 100 patients total will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma, AJCC stage IV
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as =/>20 mm with conventional techniques or as =/>10 mm with spiral CT scan. See Section 11 for the evaluation of measurable disease. Measurable disease must be present outside a previous radiation field or if inside, it must be a new lesion.
3. At least 6 months must have elapsed after completion of adjuvant therapy (if applicable).
4. Age =/>18 years.
5. ECOG Performance Status 0-1 (Karnofsky =/>60%).
6. Patients must have adequate organ and marrow function as defined below: 1) leukocytes =/>3,000 cells/mm^3; 2) absolute neutrophil count =/>1,500 cells/mm^3; 4) platelets =/>100,000 cells/mm^3; 5) total bilirubin <1.5mg/dl; 6) AST(SGOT)/ALT(SGPT) =/<2.5 X institutional upper limit of normal for patients without liver metastasis, =/< 5X institutional upper limit of normal for patients with liver metastasis; 7) creatinine - within normal institutional limits OR creatinine clearance =/>60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
7. Fasting blood glucose =/<160 mg/dl, prior to study enrollment. (For higher values, blood glucose may be controlled by dietary intervention, oral hypoglycemics and/ or insulin prior to enrollment).
8. Women of child-bearing potential (defined as not post-menopausal for 12 months or no previous surgical sterilization) and fertile men must agree to use adequate contraception for the duration of study participation. Acceptable contraception is defined as double-barrier methods (any double combination of: IUD, male or female condom with spermicidal gel, diaphragm, sponge, cervical cap). Acceptable contraception must be used for 90 days after last dose of study drugs.
9. (Continuation of inclusion criteria # 8) Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
10. Ability to understand and the willingness to sign a written informed consent document. Signed informed consent form must be obtained prior to initiation of study evaluations and/or activities.
11. INR <1.5 (or =/<3 if on anticoagulation therapy)
12. Both men and women and members of all races and ethnic groups are eligible for this trial.
13. In phase II expansion cohort, which is primarily for predictive biomarker correlation, patients enrolled will be those with pre-existing core biopsies of primary tumor or metastatic site or must be willing to undergo a biopsy for correlative studies.

Exclusion Criteria:

1. Prior systemic chemotherapy or biological therapy for metastatic disease
2. Prior exposure to IGF-1R inhibitors.
3. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the agents used in the study.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Pregnant or nursing women are excluded from this study because there is an unknown but potential risk for adverse events in infants secondary to treatment of the mother the study agents. If a pregnancy test (serum or urine) is positive, patient will be excluded.
7. Patients who are known to be HIV-positive are ineligible because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
8. No other prior malignancy is allowed except for the following: adequately treated basal or squamous cell skin cancer, in situ cervical cancer, or any other cancer from which the patient has been disease-free for two years.
9. Patients must not be currently enrolled in a therapeutic study for pancreatic cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-11-13 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milind Javle, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Abdel-Wahab R, Varadhachary GR, Bhosale PR, Wang X, Fogelman DR, Shroff RT, Overman MJ, Wolff RA, Javle M. Randomized, phase I/II study of gemcitabine plus IGF-1R antagonist (MK-0646) versus gemcitabine plus erlotinib with and without MK-0646 for advanced pancreatic adenocarcinoma. J Hematol Oncol. 2018 May 30;11(1):71. doi: 10.1186/s13045-018-0616-2. PMID 29843755
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Completed, last patient enrolled in September 26th, 2013
Groups:
- Arm A / Phase I: Arm A: MK-0646 (MK) + gemcitabine (G) G dose: 1000 mg/m2 over 100 min on D1,8,15 of a 28-day cycle MK dose: intravenously at two dose levels: 5 mg/kg (level I) or 10 mg/kg (level II) on D1,8,15,22.
- Arm B / Phase I: Arm B: MK-0646 (MK) + gemcitabine (G) + Erolotinib (E) G dose: 1000 mg/m2 over 100 min on D1,8,15 of a 28-day cycle E dose: 100 mg orally daily MK dose: intravenously at two dose levels: 5 mg/kg (level I) or 10 mg/kg (level II) on D1,8,15,22.
- Arm A / Phase II Randomization: Arm A: MK-0646 (MK) + gemcitabine (G) G dose: 1000 mg/m2 over 100 min on D1,8,15 of a 28-day cycle MK dose: 10 mg/kg
- Arm B / Phase II Randomization: Arm B: MK-0646 (MK) + gemcitabine (G) + Erolotinib (E) G dose: 1000 mg/m2 over 100 min on D1,8,15 of a 28-day cycle E dose: 100 mg orally daily MK dose: 5 mg/kg
- Arm C / Phase II Randomization: Arm C: gemcitabine (G) + Erolotinib (E) G dose: 1000 mg/m2 over 100 min on D1,8,15 of a 28-day cycle E dose: 100 mg orally daily
- Phase II Expansion: MK-0646 (MK) + gemcitabine (G) G dose: 1000 mg/m2 over 100 min on D1,8,15 of a 28-day cycle MK dose: 10 mg/kg
Period: Overall Study
Arm/Group | Arm A / Phase I | Arm B / Phase I | Arm A / Phase II Randomization | Arm B / Phase II Randomization | Arm C / Phase II Randomization | Phase II Expansion
Started | 9 | 13 | 15 | 15 | 16 | 9
Completed | 9 | 12 | 15 | 15 | 15 | 9
Not Completed | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A / Phase I: Arm A: MK-0646 (MK) + gemcitabine(G) G dose: 1000 mg/m2 over 100 min on D1,8,15 of a 28-day cycle MK dose: intravenously at two dose levels: 5 mg/kg (level I) or 10 mg/kg (level II) on D1,8,15,22. .
- Total: Total of all reporting groups
Arm/Group | Arm A / Phase I | Arm B / Phase I | Arm A / Phase II Randomization | Arm B / Phase II Randomization | Arm C / Phase II Randomization | Phase II Expansion | Total
Number analyzed (Participants) | 9 | 12 | 15 | 15 | 15 | 9 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 9 | 10 | 7 | 6 | 42
  >=65 years | 4 | 7 | 6 | 5 | 8 | 3 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.56 (7.21) | 63.33 (12.57) | 62.33 (7.66) | 62.27 (7.62) | 67.8 (8.41) | 60.89 (9.43) | 63.5 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 7 | 6 | 5 | 4 | 28
  Male | 6 | 9 | 8 | 9 | 10 | 5 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 3 | 0 | 4
  Not Hispanic or Latino | 9 | 11 | 15 | 14 | 12 | 8 | 69
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 1 | 0 | 1 | 4
  White | 9 | 10 | 12 | 13 | 10 | 7 | 61
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 3 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 9 | 12 | 15 | 15 | 15 | 9 | 75

OUTCOME MEASURES:

1. Primary Outcome: MK-0646 Maximum Tolerable Dose
Description: MK-0646 10 mg/kg was declared to be the MTD in combination with gemcitabine and 5 mg/kg the MTD in combination with Gemcitabine and erlotinib
Time Frame: up to 12 cycles
Population: The primary endpoint is MTD which was analyzed based on phase I participants only. Phase II (Arms A and B) or phase II expansion participants were not included in the analysis per design.
Measure: Number; unit: participants
Arm/Group | Arm A / Phase I | Arm B / Phase I | Arm A / Phase II Randomization | Arm B / Phase II Randomization | Arm C / Phase II Randomization | Phase II Expansion
Number analyzed (Participants) | 9 | 12 | 0 | 0 | 0 | 0
participants
  MK 5mg +G: #DLT: number analyzed (Participants) | 3 | 6 | 0 | 0 | 0 | 0
  MK 5mg +G: #DLT | 0 | 0 |  |  |  |
  MK 10mg +G: # DLT: number analyzed (Participants) | 6 | 6 | 0 | 0 | 0 | 0
  MK 10mg +G: # DLT | 0 | 2 |  |  |  |

2. Primary Outcome: Progression Free Survival
Description: Time interval (in months) from date of randomization until the date of first documented progression or date of death from any cause, whichever came first
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Population: For any group that was not analyzed for Progression Free Survival (PFS) outcome the number of participants has been set to be zero.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm B / Phase II Randomization: Arm B: MK-0646 (MK) + gemcitabine (G) + Erolotinib (E)G dose: 1000 mg/m2 over 100 min on D1,8,15 of a 28-day cycle E dose: 100 mg orally daily MK dose: 5 mg/kg
Arm/Group | Arm A / Phase I | Arm B / Phase I | Arm A / Phase II Randomization | Arm B / Phase II Randomization | Arm C / Phase II Randomization | Phase II Expansion
Number analyzed (Participants) | 0 | 0 | 15 | 15 | 15 | 9
months |  |  | 1.8 [1.8 to 9.7] | 1.8 [1.7 to 5.5] | 1.9 [1.8 to 5.4] | 2.0 [1.8 to NA] — Not estimable for the upper bound of the 95% CI

3. Secondary Outcome: Overall Survival
Description: Time interval (in months) from date of randomization until the date of death from any cause
Time Frame: From date of randomization until the date of death from any cause, assessed up to 100 months
Population: For any group that was not analyzed for Overall Survival (OS) outcome the number of participants has been set to be zero.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A / Phase I | Arm B / Phase I | Arm A / Phase II Randomization | Arm B / Phase II Randomization | Arm C / Phase II Randomization | Phase II Expansion
Number analyzed (Participants) | 0 | 0 | 15 | 15 | 15 | 9
months |  |  | 10.4 [3.9 to 18.9] | 7.1 [5.2 to 20.0] | 5.7 [4.0 to 9.5] | 8.2 [5.3 to NA] — Not estimable for the upper bound of the 95% CI

4. Secondary Outcome: Overall Response Rate
Description: Complete response + Partial response using RECIST (Response Evaluation Criteria in Solid Tumors)
Time Frame: From start of the treatment until disease progression/recurrence; or through study completion (average of 1 year)
Population: For any group that was not analyzed for Overall Response Rate outcome the number of participants has been set to be zero.
Measure: Count of Participants; unit: Participants
Groups:
- Arm B / Phase I: Arm B: MK-0646 (MK) + gemcitabine (G) + Erolotinib (E)G dose: 1000 mg/m2 over 100 min on D1,8,15 of a 28-day cycle E dose: 100 mg orally daily MK dose: intravenously at two dose levels: 5 mg/kg (level I) or 10 mg/kg (level II) on D1,8,15,22.
Arm/Group | Arm A / Phase I | Arm B / Phase I | Arm A / Phase II Randomization | Arm B / Phase II Randomization | Arm C / Phase II Randomization | Phase II Expansion
Number analyzed (Participants) | 0 | 0 | 15 | 15 | 15 | 9
Participants | 0 | 0 | 2 | 1 | 2 | 0

5. Secondary Outcome: Treatment Toxicity
Description: Number of patients who developed toxicity from treatment according to the National Cancer Institute's Common Terminology Criteria
Time Frame: Through the treatment cycles
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A / Phase I | Arm B / Phase I | Arm A / Phase II Randomization | Arm B / Phase II Randomization | Arm C / Phase II Randomization | Phase II Expansion
Number analyzed (Participants) | 9 | 12 | 15 | 15 | 15 | 9
Participants | 9 | 12 | 15 | 15 | 15 | 9

6. Other Pre Specified Outcome: Correlation Between Tissue IGF-I Expression in Patients Treated With MK-0646 and OS
Description: IGF1 expression in tissue was measured and correlated with 1 year patients survival. Inadequate biopsy data for outcome measure.
Time Frame: After completing treatment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Correlation Between Plasma IGF-I Expression in Patients Treated With MK-0646 and OS
Description: IGF1 expression in plasma was measured in patients and correlated with 1 year patients survival.
  Inadequate biopsy data for outcome measure.
Time Frame: After completing treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: assessed up to 100 months
Arm/Group | Arm A / Phase I | Arm B / Phase I | Arm A / Phase II Randomization | Arm B / Phase II Randomization | Arm C / Phase II Randomization | Phase II Expansion
All-Cause Mortality (participants affected / at risk) | 9/9 | 12/12 | 15/15 | 15/15 | 15/15 | 9/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 2/12 | 2/15 | 4/15 | 1/15 | 1/9
Other Adverse Events (participants affected / at risk) | 9/9 | 12/12 | 15/15 | 15/15 | 12/15 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A / Phase I (N=9) | Arm B / Phase I (N=12) | Arm A / Phase II Randomization (N=15) | Arm B / Phase II Randomization (N=15) | Arm C / Phase II Randomization (N=15) | Phase II Expansion (N=9)
G4 thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1 | 0
G4 neutropenia for ≥7 days (Blood and lymphatic system disorders) | 0 | 2 | 2 | 4 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A / Phase I (N=9) | Arm B / Phase I (N=12) | Arm A / Phase II Randomization (N=15) | Arm B / Phase II Randomization (N=15) | Arm C / Phase II Randomization (N=15) | Phase II Expansion (N=9)
Anemia (Blood and lymphatic system disorders) | 7 | 5 | 7 | 4 | 9 | 1
Leukopenia (Blood and lymphatic system disorders) | 9 | 10 | 6 | 4 | 5 | 0
Neutropenia (Blood and lymphatic system disorders) | 9 | 8 | 6 | 7 | 9 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 7 | 9 | 8 | 11 | 7
Lymphopenia (Blood and lymphatic system disorders) | 7 | 3 | 3 | 0 | 3 | 1
Fatigue (General disorders) | 6 | 10 | 6 | 4 | 7 | 8
Elevated ALK (Hepatobiliary disorders) | 3 | 3 | 5 | 1 | 2 | 0
Elevated ALT (Hepatobiliary disorders) | 4 | 6 | 5 | 3 | 2 | 3
Elevated AST (Hepatobiliary disorders) | 5 | 5 | 6 | 6 | 3 | 2
Elevated INR (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalemia (Investigations) | 1 | 0 | 1 | 1 | 1 | 0
Hyponatremia (Investigations) | 2 | 3 | 2 | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Other cardiac toxicity (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycemia (Endocrine disorders) | 7 | 6 | 8 | 5 | 2 | 2
Anorexia (Gastrointestinal disorders) | 3 | 6 | 2 | 4 | 5 | 1
Nausea (Gastrointestinal disorders) | 4 | 7 | 2 | 3 | 7 | 4
GIT hemorrhage (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 6 | 1 | 7 | 5 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0
Pulmonary embolism (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0
Infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT00769483/Prot_SAP_000.pdf